CLINICAL TRIAL: NCT03606174
Title: A Phase 2 Study of Sitravatinib in Combination With PD-(L)1 Checkpoint Inhibitor Regimens in Patients With Advanced or Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to sponsor decision / portfolio prioritization, and not due to safety reasons.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 516-003
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Urothelial Carcinoma; Urothelial Carcinoma Bladder; Urothelial Carcinoma Ureter; Urothelial Carcinoma of the Renal Pelvis and Ureter; Urothelial Carcinoma Urethra
Keywords: MGCD516; Antineoplastic Agents; Immunologic Factors; Nivolumab; Tyrosine Kinase Inhibitor; VEGFR; TAM RTKs; PD-1; PD-L1; Pembrolizumab; Enfortumab vedotin; Checkpoint Inhibitors; Antibody Drug Conjugates; ADC
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — sitravatinib; Nivolumab; pembrolizumab; enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: There are 9 cohorts (having 9-55 maximum patients enrolled in each; based upon response rate). Patients are assigned to cohorts based upon their prior treatments for urothelial carcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Patients previously treated with checkpoint inhibitor and platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 2 (Experimental): Patients previously treated with checkpoint inhibitor, but ineligible for platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 3 (Experimental): Patients previously treated with selected immunotherapies and platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 4 (Experimental): Patients previously treated with with selected immunotherapies, but ineligible for platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 5 (Experimental): Patients previously treated with platinum-based chemotherapy, but never treated with checkpoint inhibitor. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 6 (Experimental): Patients ineligible for treatment with platinum-based chemotherapy and never treated with checkpoint inhibitor. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 7 (Experimental): Patients previously treated with antibody-drug conjugate, checkpoint inhibitor and platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 8 (Experimental): Patients previously treated with antibody-drug conjugate and checkpoint inhibitor, but ineligible for platinum-based chemotherapy. Nivolumab over 30 min IV infusion (240 mg IV every 2 weeks or 480 mg every 4 weeks) and sitravatinib 120 mg orally once per day continuously in 28-day cycles.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Cohort 9 (Experimental): Patients previously treated with checkpoint inhibitor and platinum-based chemotherapy. There are 2 parts to this Cohort - a lead-in dose escalation portion and a dose expansion portion. In the dose escalation portion, treatment with up to 3 dose levels of sitravatinib in combination with up to 2 dose levels of pembrolizumab and enfortumab combination regimen to determine the recommended doses to be used in the combination treatment regimen and those doses will be further studied in the dose expansion portion. Pembrolizumab 200 mg over 30 min IV infusion every 3 weeks, sitravatinib orally once per day continuously in 21-day cycles (at 35 mg, 50 mg, 70 mg, or 100 mg) and enfortumab vedotin over 30 min IV infusion on Day 1 and Day 8 in 21-day cycles (at 1 mg/kg or 1.25 mg/kg).
  Interventions: Drug: Sitravatinib; Drug: Pembrolizumab; Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases
  Other Names: MGCD516
Drug: Nivolumab — Nivolumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: Opdivo
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Cohort 8
Drug: Pembrolizumab — Pembrolizumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: Keytruda
  Arms: Cohort 9
Drug: Enfortumab vedotin — Enfortumab is a Nectin-4 directed antibody-drug conjugate (ADC) comprised of a monoclonal antibody conjugated to the small molecule microtubule disrupting agent, monomethyl auristatin E (MMAE)
  Other Names: Padcev
  Arms: Cohort 9

SUMMARY:
The study will evaluate the clinical activity of PD-(L)1 Checkpoint Inhibitor regimens in combination with the investigational agent sitravatinib in patients with advanced or metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
Sitravatinib is an orally-available, small molecule inhibitor of a closely related spectrum of receptor tyrosine kinases (RTKs) including MET, Axl, MERTK, VEGFR family, PDGFR family, KIT, FLT3, Trk family, RET, DDR2 and selected Eph family members. Nivolumab is a human IgG monoclonal antibody that binds to the programmed cell death-1(PD-1) receptor and blocks its interaction with programmed cell death ligand-1 (PD-L1) and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response including anti-tumor immune response. Combining an immunotherapeutic PD-L1 checkpoint inhibitor with an agent that has both immune modulatory and antitumor properties could enhance the antitumor efficacy observed with either agent alone. Sitravatinib selectively inhibits key molecular and cellular pathways strongly implicated in checkpoint inhibitor resistance and therefore represents a rational strategy to enhance or restore anti-tumor immunity when combined with nivolumab, a checkpoint inhibitor therapy.

Pembrolizumab is a humanized IgG4 monoclonal antibody that binds to the PD-1 receptor and selectively blocks its interaction with PD-L1 and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response, including the anti-tumor immune response. Enfortumab vedotin (enfortumab) is an investigational ADC that is comprised of a fully human anti-Nectin-4 IgG1 monoclonal antibody conjugated to MMAE via a protease-cleavable linker. Enfortumab binds to cells that express Nectin-4 with high affinity, triggering the internalization and release of MMAE in target cells, inducing cell cycle arrest and apoptotic cell death. Early efficacy results from enfortumab in combination with pembrolizumab in frontline cisplatin-ineligible urothelial carcinoma in the ongoing EV-103 study have demonstrated encouraging activity with a safety profile that appears manageable and tolerable. Addition of sitravatinib to this combination might further augment clinical activity by selectively inhibiting key molecular and cellular pathways strongly implicated in checkpoint inhibitor resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of urothelial carcinoma
* Adequate bone marrow and organ function

Exclusion Criteria:

* Uncontrolled tumor in the brain
* Unacceptable toxicity with prior checkpoint inhibitor
* Impaired heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirak Der-Torossian, MD, Study Director — Mirati Therapeutics Inc.
Locations (36):
- United States (36):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California Irvine, Irvine, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - SCRI - Florida Cancer Specialists- North Region, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach, West Palm Beach, Florida
  - The University of Chicago, Chicago, Illinois
  - Indiana University - Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Norton Cancer Institute - Broadway, Louisville, Kentucky
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Maryland Oncology Hematology, P.A., Lanham, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Southwest, Las Vegas, Nevada
  - New York Oncology Hematology - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - NYU Langone Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York-Presbyterian - Weill Cornell Medical Center, New York, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University - Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology- Memorial City, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists- Fairfax, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Seattle Cancer Center Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 260 participants were enrolled into this study at investigative sites in the United States.
Pre-assignment Details: Screening tests and procedures were performed within the 28 days preceding administration of the first dose.
Groups:
- Cohort 1: Participants with locally advanced or metastatic urothelial carcinoma (UC) with documented disease progression on or after previous anti-programmed cell death (PD)-ligand(L)-1 as most recent treatment, and who were previously treated with a platinum-based chemotherapy were enrolled into Cohort 1.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules once daily (QD) in 28-day cycles. Nivolumab was received via an intravenous (IV) infusion over approximately 30 minutes (± 5 minutes) at 240 mg once every 2 weeks (Q2W) or 480 mg once every 4 weeks (Q4W), at the discretion of the Investigator and in accordance with the current nivolumab US Prescribing Information (USPI).
- Cohort 2: Participants with locally advanced or metastatic UC with documented disease progression on or after previous anti-PD-L-1 as most recent treatment, and who were considered ineligible for platinum-based chemotherapy were enrolled into Cohort 2.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 3: Participants with locally advanced or metastatic UC with documented disease progression on or after a previous anti PD-(L)1 as the most recent treatment, who previously received (in combination or separately) other selected immunotherapies, and who were previously treated with a platinum-based chemotherapy were enrolled into Cohort 3.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 4: Participants with locally advanced or metastatic UC with documented disease progression on or after a previous anti-PD-(L)1 as the most recent treatment, who previously received (in combination or separately) other selected immunotherapies, and who were considered ineligible for platinum-based chemotherapy were enrolled into Cohort 4.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 5: Participants with locally advanced or metastatic UC who had not previously received an anti-PD-(L)1, and who were previously treated with a platinum-based chemotherapy were enrolled into Cohort 5.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 6: Participants with locally advanced or metastatic UC who had not previously received an anti-PD-(L)1, and who were considered ineligible for platinum-based chemotherapy were enrolled into Cohort 6.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 120 mg capsules QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 7: Participants with locally advanced or metastatic UC with documented disease progression on or after a previous anti PD-(L)1 and antibody-drug conjugate (ADC) (in combination or separately, and in any order), and who were previously treated with a platinum-based chemotherapy were enrolled into Cohort 7.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 100 mg malate capsules, or 120 mg free base capsule formulation QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 8: Participants with locally advanced or metastatic UC with documented disease progression on or after a previous anti PD-(L)1 and ADC (in combination or separately, and in any order), and who were considered ineligible for platinum-based chemotherapy were enrolled into Cohort 8.
  Participants received sitravatinib in combination with nivolumab. Sitravatinib was received orally via 100 mg malate capsules, or 120 mg free base capsule formulation QD in 28-day cycles. Nivolumab was received via an IV infusion over approximately 30 minutes (± 5 minutes) at 240 mg Q2W or 480 mg Q4W, at the discretion of the Investigator and in accordance with the current nivolumab USPI.
- Cohort 9 Dose Level 1: Participants with locally advanced or metastatic UC who had previously received a PD-(L)1 checkpoint inhibitor (CPI) and a platinum-based chemotherapy were enrolled into Cohort 9, which included a lead-in dose-escalation part. A dose-expansion part was planned, but was not enrolled.
  During the lead-in dose-escalation part, participants in Cohort 9 Dose Level 1 were enrolled to receive sitravatinib 35 mg QD orally via capsules in 21-day cycles, enfortumab vedotin 1.25 mg/kg IV infusion on Days 1 and 8 every 3 weeks (Q3W), and pembrolizumab 200 mg Q3W as an IV infusion.
- Cohort 9 Dose Level 2: Participants with locally advanced or metastatic UC who had previously received a PD-(L)1 checkpoint inhibitor (CPI) and a platinum-based chemotherapy were enrolled into Cohort 9, which included a lead-in dose-escalation part. A dose-expansion part was planned, but was not enrolled.
  During the lead-in dose-escalation part, participants in Cohort 9 Dose Level 2 were enrolled to receive sitravatinib 35 mg QD orally via capsules in 21-day cycles, enfortumab vedotin 1.0 mg/kg IV infusion on Days 1 and 8 Q3W, and pembrolizumab 200 mg Q3W as an IV infusion.
- Cohort 9 Dose Level 3: Participants with locally advanced or metastatic UC who had previously received a PD-(L)1 checkpoint inhibitor (CPI) and a platinum-based chemotherapy were enrolled into Cohort 9, which included a lead-in dose-escalation part. A dose-expansion part was planned, but was not enrolled.
  During the lead-in dose-escalation part, participants in Cohort 9 Dose Level 3 were enrolled to receive sitravatinib 70 mg QD orally via capsules in 21-day cycles, enfortumab vedotin 1.0 mg/kg IV infusion on Days 1 and 8 Q3W, and pembrolizumab 200 mg Q3W as an IV infusion.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
Started | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4
Started Cohort 9 Lead-in Dose-escalation Part | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 8 | 4 | 4
Started Cohort 9 Dose-expansion Part | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 (N/A for Cohorts 1-8) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4
Not completed — Death | 37 | 15 | 15 | 7 | 35 | 12 | 35 | 8 | 5 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 5 | 7 | 3 | 0 | 11 | 6 | 12 | 1 | 3 | 1 | 2
Not completed — Miscellaneous | 1 | 1 | 0 | 1 | 4 | 7 | 5 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Measured in the safety population, which included all participants who received ≥ 1 dose of any study treatment (sitravatinib, nivolumab, pembrolizumab, or enfortumab vedotin).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3 | Total
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.63) | 72.3 (7.94) | 67.6 (12.89) | 75.1 (7.62) | 65.2 (8.34) | 70.0 (8.23) | 67.1 (9.07) | 78.0 (7.02) | 65.1 (6.40) | 69.0 (8.00) | 75.8 (9.54) | 68.3 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 6 | 1 | 10 | 10 | 17 | 4 | 0 | 1 | 1 | 70
  Male | 36 | 16 | 12 | 8 | 43 | 17 | 39 | 5 | 8 | 3 | 3 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 10
  Not Hispanic or Latino | 44 | 23 | 18 | 7 | 52 | 27 | 53 | 8 | 8 | 4 | 4 | 248
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 0 | 5 | 1 | 2 | 0 | 0 | 1 | 0 | 14
  White | 46 | 21 | 15 | 9 | 46 | 26 | 48 | 8 | 8 | 2 | 3 | 232
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the number of participants documented to have a confirmed investigator-assessed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must have decreased to normal size (short axis < 10 mm). PR was defined as a greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Up to approximately 3 years
Population: Measured in the Full Analysis Set, which included participants who received ≥ 1 dose of each study treatment drug (ie, ≥ 1 dose of both sitravatinib and nivolumab for Cohorts 1 to 8, or ≥ 1 dose each of sitravatinib, pembrolizumab, and enfortumab vedotin for Cohort 9). Per the statistical analysis plan (SAP), Cohort 9 arms are grouped as pre-specified as there was never intent to compare efficacy endpoints across Cohort 9 dose levels.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 9: Participants with locally advanced or metastatic UC who had previously received a PD-(L)1 checkpoint inhibitor (CPI) and a platinum-based chemotherapy were enrolled into Cohort 9, which included a lead-in dose-escalation part. A dose-expansion part was planned, but was not enrolled.
  During the lead-in dose-escalation part, participants were enrolled to 3 dose levels of sitravatinib in combination with pembrolizumab and enfortumab vedotin. Sitravatinib was received orally via capsules QD in 21-day cycles at doses 35 mg and 70 mg. Pembrolizumab was received as an IV infusion over approximately 30 minutes (± 5 minutes) at 200 mg every 3 weeks (Q3W), in accordance with the current pembrolizumab USPI. Enfortumab vedotin dosing was based on participant weight, starting at 1.25 mg/kg up to 125 mg/kg QD, with a dose de-escalation step to 1 mg/kg. Enfortumab vedotin was received as an IV infusion over approximately 30 minutes (± 5 minutes) on Days 1 and 8 of a 21-day cycle.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 16
Participants | 6 | 5 | 4 | 0 | 17 | 9 | 3 | 0 | 4

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any reaction, side effect or other undesirable medical event that occurred during participation in a clinical trial, regardless of treatment group or suspected causal relationship to study treatment. Any clinically significant changes from baseline in laboratory results were recorded as AEs.
Time Frame: Day 1 up to approximately 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4
Participants | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4

3. Secondary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE was defined as any event that resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/permanent damage (substantial disruption of the ability to conduct normal life functions), a congenital anomaly/birth defect, or may have jeopardized the participant and may have required medical or surgical intervention to prevent intensive treatment in an emergency room or at home (e.g. for allergic bronchospasm, blood dyscrasias or convulsions) that do not result in inpatient hospitalization, development of drug dependency or drug abuse.
Time Frame: Day 1 up to approximately 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4
Participants | 35 | 15 | 10 | 4 | 26 | 14 | 23 | 3 | 5 | 1 | 3

4. Secondary Outcome: Number of Participants Who Experienced a Treatment-related Adverse Event
Description: A treatment-related adverse event was defined as an adverse event determined to have a possible causal relationship to the study treatment(s) by the investigator. An adverse event was defined as any reaction, side effect or other undesirable medical event that occurred during participation in a clinical trial. Any clinically significant changes from baseline in laboratory results were recorded as adverse events.
Time Frame: Day 1 up to approximately 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 8 | 4 | 4
Participants
  Sitravatinib Related | 43 | 23 | 18 | 8 | 51 | 26 | 52 | 9 | 8 | 4 | 3
  Nivolumab Related | 41 | 23 | 15 | 7 | 41 | 24 | 35 | 4 | NA — As pre-specified, participants did not receive nivolumab treatment in this Cohort. | NA — As pre-specified, participants did not receive nivolumab treatment in this Cohort. | NA — As pre-specified, participants did not receive nivolumab treatment in this Cohort.
  Pembrolizumab Related | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | NA — As pre-specified, participants did not receive pembrolizumab treatment in this Cohort. | 6 | 3 | 3
  Enfortumab Vedotin Related | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | NA — As pre-specified, participants did not receive enfortumab vedotin treatment in this Cohort. | 7 | 4 | 4

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of objective progression of disease (PD) per RECIST V1.1, or to death due to any cause in the absence of documented PD. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must have decreased to normal size (short axis < 10 mm). PR was defined as a greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
  Per the statistical analysis plan (SAP), Cohort 9 arms are grouped as pre-specified as there was never intent to compare efficacy endpoints across Cohort 9 dose levels.
Time Frame: Up to approximately 3 years
Population: Measured in the Clinical Activity Evaluable Population-confirmed Response Subset, which included participants who achieved an objective response, received ≥1 dose of study treatment drug, had an evaluable baseline tumor assessment and ≥1 post-baseline tumor assessment. One participant in Cohort 6 who experienced a response wasn't included in DOR analysis because they didn't receive ≥1 dose of study treatment, have an evaluable baseline tumor assessment or ≥1 post-baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 6 | 5 | 4 | 0 | 17 | 8 | 3 | 0 | 4
months | 5.585 [3.844 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response. | 9.478 [5.782 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response. | 11.762 [7.392 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response. |  | 7.326 [5.520 to 12.977] | 16.361 [5.552 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response. | 7.425 [5.552 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response. |  | 11.8 [4.70 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a response.

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) was defined as the number of participants documented to have a confirmed CR, PR, or stable disease (SD), per RECIST V1.1, documented during at least 1 on-study assessment. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must have decreased to normal size (short axis < 10 mm). PR was defined as a greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. SD was defined as target lesions increasing by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer holds.
Time Frame: Up to approximately 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 16
Participants | 32 | 19 | 12 | 7 | 35 | 17 | 33 | 6 | 10

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first study treatment to first PD per RECIST V1.1, or death due to any cause in the absence of documented PD.
Time Frame: Up to approximately 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 16
months | 3.877 [2.497 to 5.487] | 7.786 [3.943 to 14.620] | 3.910 [1.873 to 9.133] | 3.515 [1.971 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a documented PD or death. | 3.943 [3.450 to 5.651] | 5.421 [3.220 to 18.168] | 3.680 [2.234 to 5.520] | 3.713 [1.840 to NA] — Upper confidence intervals could not be calculated due to the low number of participants with a documented PD or death. | 4.0 [2.04 to 6.51]

8. Secondary Outcome: 1-Year Survival Rate
Description: Survival was defined as the time from date of first study treatment to death due to any cause. Kaplan-Meier (product limit) estimates of the percentage of participants who died at 1-year was calculated to estimate the 1-year survival rate, defined as the percentage of participants alive at 1 year. Confidence Intervals were calculated based on Greenwood's formula. Participants who discontinued prior to 1-year were censored on the last date that they were known to be alive. For participants with no follow-up after first dose of study drug, survival rate was censored at the date of first dose (Day 1).
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 16
percentage of participants | 42.5 [27.9 to 56.4] | 56.5 [34.3 to 73.8] | 55.6 [30.5 to 74.8] | 44.4 [13.6 to 71.9] | 53.9 [39.5 to 66.3] | 57.1 [36.0 to 73.6] | 32.6 [19.5 to 46.3] | 16.7 [1.1 to 49.3] | 41.5 [15.4 to 66.1]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of first study treatment to death due to any cause.
Time Frame: Up to approximately 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 18 | 9 | 53 | 27 | 56 | 9 | 16
months | 8.049 [4.632 to 15.967] | 15.639 [7.655 to NA] — Data could not be calculated as too few participants experienced an event. | 12.945 [5.618 to 22.439] | 5.092 [1.971 to 24.279] | 13.405 [5.782 to 21.290] | NA [5.947 to NA] — Data could not be calculated as too few participants experienced an event. | 8.969 [7.359 to 10.809] | 7.556 [2.825 to 9.922] | 10.8 [2.69 to NA] — Data could not be calculated as too few participants experienced an event.

10. Secondary Outcome: Geometric Mean Blood Plasma Concentration of Sitravatinib
Description: Blood draws for analysis of blood plasma concentrations of sitravatinib were collected following electrocardiograms and assessment of vital signs. Concentration data below the limit of quantification were set to 0.
Time Frame: Cycle(C)1 Day(D)1 pre-dose, 30min, 2,4,6,7,8,24hr post-dose, C1D15 pre-dose, 30min,2,4,6,7,8,24hr post-dose, C2D1 pre-dose,7hr post-dose, C2D8,C3D1,C3D8,C5D1,C6D8 pre-dose (28 day cycles Cohorts 1-8, 21 day cycles Cohort 9)
Population: Measured in the Pharmacokinetic (PK) Evaluable Population, which included all participants who received treatment with sitravatinib and had available data at each timepoint. Per the statistical analysis plan (SAP), Cohort 9 arms are grouped as pre-specified as there was never intent to compare PK endpoints across Cohort 9 dose levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9
Number analyzed (Participants) | 49 | 23 | 17 | 9 | 53 | 27 | 56 | 9 | 16
ng/mL
  Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 46 | 21 | 16 | 9 | 50 | 24 | 46 | 8 | 16
  Cycle 1 Day 1 Pre-dose | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 1 30 Min Post-Dose: number analyzed (Participants) | 34 | 15 | 15 | 6 | 41 | 18 | 42 | 7 | 12
  Cycle 1 Day 1 30 Min Post-Dose | 1.85 (300.88) | 0.82 (10.95) | 1.56 (176.68) | 0.91 (499.94) | 1.25 (266.58) | 1.28 (231.33) | 1.40 (268.79) | 0.25 (248.74) | 0.40 (172.86)
  Cycle 1 Day 1 2 Hours Post-Dose: number analyzed (Participants) | 7 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 2 Hours Post-Dose | 5.69 (117.10) |  | 6.94 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  | 24.90 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 1 4 Hours Post-Dose: number analyzed (Participants) | 44 | 12 | 10 | 5 | 26 | 0 | 1 | 0 | 0
  Cycle 1 Day 1 4 Hours Post-Dose | 16.55 (168.43) | 21.46 (122.57) | 31.21 (80.61) | 18.33 (158.02) | 23.72 (104.51) |  | 35.20 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |
  Cycle 1 Day 1 6 Hours Post-Dose: number analyzed (Participants) | 7 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 6 Hours Post-Dose | 23.16 (69.50) |  | 11.70 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  | 15.50 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 1 7 Hours Post-Dose: number analyzed (Participants) | 1 | 6 | 2 | 4 | 13 | 7 | 21 | 5 | 11
  Cycle 1 Day 1 7 Hours Post-Dose | 27.40 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. | 22.90 (121.87) | 20.08 (167.73) | 15.36 (108.29) | 23.13 (167.10) | 23.13 (126.44) | 37.99 (50.79) | 31.21 (39.99) | 10.56 (41.43)
  Cycle 1 Day 1 8 Hours Post-Dose: number analyzed (Participants) | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 8 Hours Post-Dose | 26.08 (72.20) |  | 12.10 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  | 23.00 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 1 24 Hours Post-Dose: number analyzed (Participants) | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 24 Hours Post-Dose | 24.82 (71.41) |  |  |  | 26.30 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 15 Pre-Dose: number analyzed (Participants) | 37 | 15 | 12 | 8 | 34 | 9 | 34 | 4 | 0
  Cycle 1 Day 15 Pre-Dose | 66.00 (52.30) | 50.21 (92.49) | 42.03 (232.08) | 55.22 (34.39) | 50.58 (51.48) | 70.11 (67.12) | 49.94 (60.28) | 47.01 (39.78) |
  Cycle 1 Day 15 30 Min Post-Dose: number analyzed (Participants) | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 30 Min Post-Dose | 54.47 (77.06) |  |  |  | 75.00 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 15 2 Hours Post-Dose: number analyzed (Participants) | 8 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 2 Hours Post-Dose | 62.50 (44.94) |  |  |  | 67.80 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 15 4 Hours Post-Dose: number analyzed (Participants) | 34 | 7 | 10 | 4 | 21 | 3 | 2 | 1 | 0
  Cycle 1 Day 15 4 Hours Post-Dose | 70.90 (49.99) | 68.77 (23.87) | 52.36 (111.45) | 95.35 (3.65) | 68.67 (52.79) | 45.27 (21.03) | 50.71 (33.36) | 55.30 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |
  Cycle 1 Day 15 6 Hours Post-Dose: number analyzed (Participants) | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 6 Hours Post-Dose | 67.45 (55.03) |  |  |  | 82.90 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 15 7 Hours Post-Dose: number analyzed (Participants) | 0 | 3 | 2 | 4 | 9 | 3 | 19 | 2 | 0
  Cycle 1 Day 15 7 Hours Post-Dose |  | 89.19 (10.73) | 81.09 (85.63) | 62.78 (22.36) | 75.08 (45.43) | 104.61 (26.97) | 76.70 (51.05) | 86.04 (2.22) |
  Cycle 1 Day 15 8 Hours Post-Dose: number analyzed (Participants) | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 8 Hours Post-Dose | 72.12 (58.96) |  |  |  | 95.20 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 1 Day 15 24 Hours Post-Dose: number analyzed (Participants) | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 24 Hours Post-Dose | 59.88 (52.20) |  |  |  | 85.20 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable PK samples at this time point. |  |  |  |
  Cycle 2 Day 1 Pre-Dose: number analyzed (Participants) | 31 | 17 | 16 | 7 | 33 | 19 | 34 | 6 | 11
  Cycle 2 Day 1 Pre-Dose | 28.06 (184.46) | 36.81 (107.98) | 27.15 (459.38) | 48.24 (19.63) | 39.39 (101.75) | 32.81 (156.63) | 32.38 (155.83) | 46.89 (30.61) | 8.15 (274.13)
  Cycle 2 Day 1 7 Hours Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Cycle 2 Day 1 7 Hours Post-Dose |  |  |  |  |  |  |  |  | 26.28 (68.42)
  Cycle 2 Day 8 Pre-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Cycle 2 Day 8 Pre-Dose |  |  |  |  |  |  |  |  | 12.43 (476.36)
  Cycle 3 Day 1 Pre-Dose: number analyzed (Participants) | 23 | 15 | 8 | 4 | 25 | 12 | 30 | 5 | 0
  Cycle 3 Day 1 Pre-Dose | 29.10 (190.09) | 37.99 (126.82) | 32.32 (56.61) | 56.40 (45.32) | 39.28 (48.02) | 20.02 (422.49) | 29.21 (140.39) | 19.39 (259.86) |
  Cycle 3 Day 8 Pre-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Cycle 3 Day 8 Pre-Dose |  |  |  |  |  |  |  |  | 7.53 (823.64)
  Cycle 5 Day 1 Pre-Dose: number analyzed (Participants) | 16 | 9 | 8 | 3 | 18 | 10 | 23 | 2 | 0
  Cycle 5 Day 1 Pre-Dose | 33.41 (41.39) | 40.39 (20.19) | 44.45 (42.23) | 28.04 (81.00) | 26.48 (121.54) | 42.98 (39.16) | 37.55 (47.23) | 38.47 (20.17) |
  Cycle 6 Day 8 Pre-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Cycle 6 Day 8 Pre-Dose |  |  |  |  |  |  |  |  | 17.87 (105.74)

11. Secondary Outcome: Cohort 9 Lead-in Dose Escalation Part Only: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: A DLT was defined as any of the following events considered to be causally related to treatment with sitravatinib in combination with pembrolizumab and enfortumab in the lead-in dose escalation part of Cohort 9 (as pre-specified): hematological DLTs (Grade 4 neutropenia, thrombocytopenia, anemia unexplained by underlying disease, ≥Grade 3 febrile neutropenia or neutropenia with significant clinical sequelae, or any requirement for a platelet transfusion), non-hematological DLTs (≥Grade 4 infusion related reaction, non-hematological toxicity, Grade 3 infusion related reaction that does not resolve within 24 hours, hypertension that cannot be controlled with medical therapy), other Grade 3 non-hematologic toxicity lasting for >3 days, with exceptions, Grade 2 pneumonitis or colitis, ≥Grade 3 non-hematological laboratory abnormalities, alanine transaminase>3 x upper limit of normal (ULN) with bilirubin> 2xULN, and other related toxic effects may have been assessed as DLTs.
Time Frame: Cycle 1 Day 1 through pre-dose Cycle 2 Day 1 (cycle for Cohort 9 was 21 days)
Population: Measured in the DLT evaluable population, which, as pre-specified in the statistical analysis plan, was defined as participants who enrolled in the lead-in dose escalation portion of Cohort 9, who experienced a DLT or who cleared the DLT period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
Number analyzed (Participants) | 8 | 4 | 4
Participants | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 3 years
Description: All cause mortality, serious adverse events and other adverse events are reported for all enrolled participants.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 Dose Level 1 | Cohort 9 Dose Level 2 | Cohort 9 Dose Level 3
All-Cause Mortality (participants affected / at risk) | 37/49 | 15/23 | 15/18 | 7/9 | 35/53 | 12/27 | 36/56 | 8/9 | 5/8 | 3/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 35/49 | 15/23 | 10/18 | 4/9 | 26/53 | 14/27 | 23/56 | 3/9 | 5/8 | 1/4 | 3/4
Other Adverse Events (participants affected / at risk) | 49/49 | 23/23 | 18/18 | 9/9 | 53/53 | 27/27 | 56/56 | 9/9 | 8/8 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=49) | Cohort 2 (N=23) | Cohort 3 (N=18) | Cohort 4 (N=9) | Cohort 5 (N=53) | Cohort 6 (N=27) | Cohort 7 (N=56) | Cohort 8 (N=9) | Cohort 9 Dose Level 1 (N=8) | Cohort 9 Dose Level 2 (N=4) | Cohort 9 Dose Level 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=49) | Cohort 2 (N=23) | Cohort 3 (N=18) | Cohort 4 (N=9) | Cohort 5 (N=53) | Cohort 6 (N=27) | Cohort 7 (N=56) | Cohort 8 (N=9) | Cohort 9 Dose Level 1 (N=8) | Cohort 9 Dose Level 2 (N=4) | Cohort 9 Dose Level 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 13 (27) | 10 (14) | 2 (4) | 2 (3) | 10 (21) | 10 (27) | 10 (18) | 1 (2) | 2 (3) | 1 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogonadism male (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 19 (20) | 9 (9) | 8 (9) | 4 (4) | 14 (15) | 8 (9) | 13 (14) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid margin crusting (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleral discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 4 (6) | 8 (10) | 1 (1) | 9 (13) | 12 (16) | 6 (8) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (20) | 9 (10) | 5 (7) | 0 (0) | 17 (26) | 12 (16) | 17 (18) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 29 (66) | 20 (52) | 13 (24) | 4 (12) | 34 (109) | 18 (33) | 31 (66) | 3 (11) | 4 (7) | 3 (4) | 1 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 6 (7) | 3 (3) | 2 (2) | 4 (4) | 6 (7) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 3 (4) | 3 (4) | 0 (0) | 5 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 20 (37) | 12 (18) | 7 (9) | 3 (3) | 19 (26) | 13 (18) | 17 (23) | 5 (6) | 2 (7) | 3 (4) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 6 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 11 (19) | 4 (7) | 7 (9) | 2 (2) | 7 (11) | 7 (12) | 10 (18) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (23) | 7 (9) | 2 (2) | 1 (1) | 16 (22) | 7 (12) | 11 (14) | 4 (5) | 1 (3) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 35 (67) | 19 (46) | 15 (28) | 4 (5) | 32 (54) | 17 (27) | 24 (33) | 1 (1) | 3 (7) | 3 (11) | 2 (7)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (5) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 4 (4) | 1 (1) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 13 (14) | 9 (15) | 2 (2) | 1 (1) | 7 (7) | 4 (7) | 5 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 6 (7) | 2 (2) | 1 (1) | 5 (7) | 3 (4) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 3 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (16) | 8 (13) | 4 (5) | 1 (1) | 8 (14) | 6 (7) | 7 (10) | 3 (5) | 1 (1) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 4 (5) | 0 (0) | 2 (3) | 6 (7) | 6 (8) | 2 (4) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (22) | 8 (14) | 3 (3) | 2 (3) | 23 (40) | 14 (23) | 15 (16) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 10 (15) | 5 (5) | 3 (3) | 2 (3) | 3 (7) | 6 (17) | 4 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 14 (19) | 9 (11) | 5 (5) | 2 (2) | 18 (26) | 14 (32) | 17 (18) | 1 (1) | 3 (8) | 2 (2) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (9) | 5 (13) | 3 (3) | 0 (0) | 8 (10) | 6 (7) | 6 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 10 (21) | 9 (10) | 2 (2) | 1 (1) | 17 (27) | 8 (13) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 8 (9) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 10 (22) | 6 (7) | 5 (9) | 2 (6) | 6 (13) | 6 (24) | 10 (14) | 1 (2) | 1 (5) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (6) | 4 (7) | 3 (5) | 1 (2) | 5 (8) | 3 (6) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (7) | 3 (5) | 4 (10) | 1 (1) | 7 (10) | 3 (3) | 3 (3) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 15 (25) | 13 (20) | 4 (10) | 2 (2) | 14 (26) | 11 (15) | 12 (14) | 0 (0) | 2 (3) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 23 (41) | 18 (26) | 12 (21) | 3 (3) | 32 (51) | 14 (18) | 17 (24) | 1 (1) | 2 (4) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 1 (1) | 2 (2) | 8 (9) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (9) | 3 (7) | 2 (7) | 1 (1) | 4 (5) | 7 (14) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (11) | 3 (4) | 1 (2) | 1 (4) | 5 (8) | 6 (7) | 2 (2) | 3 (6) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (6) | 3 (5) | 2 (2) | 2 (2) | 7 (8) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (14) | 7 (10) | 3 (6) | 2 (3) | 8 (11) | 8 (9) | 5 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 8 (9) | 4 (4) | 4 (11) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8) | 4 (7) | 1 (4) | 2 (2) | 8 (10) | 3 (3) | 6 (13) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (12) | 4 (6) | 5 (10) | 2 (2) | 16 (29) | 7 (10) | 8 (10) | 3 (5) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (16) | 3 (4) | 1 (2) | 1 (1) | 10 (14) | 3 (3) | 11 (14) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7) | 4 (7) | 1 (1) | 11 (13) | 5 (6) | 8 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (12) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 7 (18) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 6 (8) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (7) | 3 (3) | 1 (1) | 5 (13) | 3 (3) | 2 (2) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (11) | 6 (9) | 0 (0) | 1 (1) | 14 (16) | 12 (12) | 11 (11) | 2 (2) | 3 (5) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 10 (18) | 5 (5) | 4 (5) | 4 (4) | 4 (4) | 5 (6) | 4 (4) | 0 (0) | 2 (4) | 2 (3) | 2 (2)
Headache (Nervous system disorders) | 8 (9) | 2 (3) | 3 (4) | 0 (0) | 9 (13) | 5 (5) | 9 (12) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (2) | 1 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 2 (3) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (6) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (11) | 6 (7) | 1 (1) | 2 (2) | 7 (7) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tangentiality (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 12 (14) | 3 (3) | 2 (2) | 2 (2) | 11 (19) | 1 (3) | 10 (15) | 2 (2) | 5 (7) | 0 (0) | 1 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (13) | 2 (3) | 1 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6) | 3 (3) | 2 (2) | 12 (16) | 7 (7) | 7 (8) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 15 (19) | 9 (10) | 4 (4) | 21 (28) | 9 (13) | 23 (23) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (11) | 4 (7) | 3 (3) | 19 (30) | 5 (5) | 7 (8) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (10) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (20) | 5 (11) | 7 (16) | 3 (4) | 13 (17) | 5 (6) | 5 (12) | 2 (6) | 0 (0) | 2 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 2 (3) | 1 (1) | 7 (7) | 3 (3) | 6 (6) | 0 (0) | 2 (3) | 1 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 3 (5) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7) | 3 (3) | 0 (0) | 11 (15) | 6 (7) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 14 (32) | 12 (19) | 6 (16) | 4 (5) | 21 (29) | 12 (15) | 27 (43) | 4 (4) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03606174/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03606174/SAP_001.pdf